CLINICAL TRIAL: NCT05833126
Title: Hepatic Arterial Infusion Chemotherapy in Combination With Atezolizumab and Bevacizumab for Second-line Treatment of Patients With Recurrent Liver Cancer After Liver Transplantation: an Open-label, Prospective, Single-center, Single-arm Clinical Study Protocol
Brief Title: Hepatic Arterial Infusion Chemotherapy in Combination With Atezolizumab and Bevacizumab for Second-line Treatment of Patients With Recurrent Liver Cancer After Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shuhong Yi (Other)
Responsible Party: Sponsor-Investigator, Shuhong Yi, Clinical Professor, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]02-116-99
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Liver Cancer After Liver Transplantation
Keywords: Atezolizumab; Bevacizumab; Hepatic arterial infusion chemotherapy
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic arterial infusion chemotherapy + Atezolizumab and bevacizumab (Experimental): Hepatic arterial infusion chemotherapy: percutaneous introduction of a standard hepatic arterial catheter through the femoral artery. FOLFOX was sequentially transfused by a fixed catheter. Drugs:FOLFOX regimen: oxaliplatin, calcium folinate, and 5-FU.
  Atezolizumab: About 3 to 7 days after HAIC treatment, when liver function is stable (TBILI<2 times the upper limit of normal), Atezolizumab therapy can be started. The dosage was 1200mg and was given intravenously for at least 1 hour, once every 3 weeks. The longest course of treatment is 24 months.
  Bevacizumab: About 3 to 7 days after HAIC treatment, when liver function is stable (TBILI<2 times the upper limit of normal), bevacizumab therapy can be started. The dosage was 15mg/kg and was given intravenously for no less than 1 hour, once every 3 weeks. The longest course of treatment is 24 months.
  Interventions: Drug: Hepatic arterial infusion chemotherapy + Atezolizumab and bevacizumab

INTERVENTIONS:
Drug: Hepatic arterial infusion chemotherapy + Atezolizumab and bevacizumab — Drug: Oxaliplatin, calcium folinate, 5-FU, Atezolizumab and bevacizumab Procedure: HAIC

SUMMARY:
For patients with recurrent liver cancer after liver transplantation, the median survival time is low and the prognosis is often poor. On the one hand, it is necessary to take into account the weakened effect of postoperative anti-rejection drugs with the use of immune checkpoint inhibitors, and on the other hand, the therapeutic effect of recurrent tumors should be taken into account. Both HAIC (hepatic arterial infusion chemotherapy) and T+A（Bevacizumab+Atezolizumab) have inhibitory effects on tumor, and we consider combining them organically to explore one that not only has a good inhibitory effect on tumor, but also better reduces the risk and degree of rejection. Therefore, in order to determine the feasibility and effectiveness of hepatic arterial infusion chemotherapy combined with Atezolizumab and Bevacizumab in the second-line treatment of patients with recurrent liver cancer after liver transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, ≤75 years old, gender unlimited;
2. hepatocellular carcinoma confirmed by pathology after liver transplantation;
3. CT and/or MRI confirmed tumor recurrence or metastasis, and the tumor recurrence and metastasis were not suitable for radical treatment such as surgical resection or ablation after multidisciplinary evaluation, and disease progression occurred after one first-line treatment regimen without immunotherapy;
4. There is at least one measurable recurrent or metastatic tumor lesion;
5. The expected survival time is more than 3 months;
6. Child-Pugh grade A and B (≤7 points);
7. Function of other vital organs: absolute neutrophil count ≥1.5×10E9/L; Platelet ≥50×10 e9 / L; Hemoglobin ≥9 g/dL; Serum albumin ≥2.8g/dL; Thyroid stimulating hormone (TSH)≤1 ULN(if TSH is abnormal, both T3 and T4 levels should be checked. If the levels of T3 and T4 were normal, the patients could be enrolled); Bilirubin ≤ 1.5x ULN; ALT and AST≤3 times ULN; Serum creatinine ≤1.5 ULN;
8. ECOG scored 0-2 points;
9. The patient fully understands and voluntarily signs the informed consent, and is willing and able to comply with the requirements of visit, treatment plan, laboratory examination and other requirements of the study schedule.

Exclusion Criteria:

1. Positive expression of PD-L1 in immunohistochemical liver biopsy (parenchymal or non-parenchymal cells of liver);
2. Allergic to bevacizumab and Atezolizumab;
3. ≥ grade II myocardial ischemia or myocardial infarction;
4. The hypertensive drugs cannot be controlled to the normal level (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg); Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg <2g/L), a history of gastrointestinal bleeding within 6 months;
5. Patients with high risk of bleeding or receiving thrombolytic or anticoagulant treatment;
6. Autoimmune diseases include systemic lupus erythematosus, rheumatoid arthritis, psoriasis, etc.;
7. The primary liver disease of liver transplantation was autoimmune hepatitis, primary biliary cirrhosis, or primary sclerosing cholangitis;
8. interstitial pneumonia and other lung diseases, poor lung function;
9. Participate in clinical trials of other experimental drugs within 4 weeks;
10. infections requiring systemic treatment;
11. human immunodeficiency virus (HIV) positive infection;
12. Other factors that may affect safety or compliance;
13. During treatment of acute rejection or within 1 month after treatment;
14. Poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Acute graft rejection rate | 3 months
  defined as the incidence of acute graft rejection after HAIC combined with T+A.
Objective Response Rate | 1 year
  defined as the treatment response assessed by mRECIST after HAIC combined with T+A treatment

SECONDARY OUTCOMES:
Overall Survival | 1 year
  defined as the time from HAIC combined with T+A treatment to patient death from any cause.
Progression-free Survival | 1 year
  defined as the time from the start of HAIC combined with T+A treatment to the onset of tumor Progression or death from any cause.
Time to Progression | 1 year
  defined as the time from the start of HAIC combined with T+A treatment to tumor progression or death from any cause.
Serious Adverse Event | 1 year
  The incidence of serious adverse events caused by HAIC combined with T+A treatment.
Graft Rejection | 1 year
  defined as the incidence of transplant rejection during HAIC combined with T+A treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhong Yi, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Liver Transplantation, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided